CLINICAL TRIAL: NCT00536523
Title: Women's Cancer Center Protocol #52: Alterations in Serum Serotonin Levels as a Mechanism for Chemotherapy Induced Constipation
Brief Title: Effect of Serotonin Level on Constipation Caused by Chemotherapy in Patients With Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Terminated | Type: Observational
Why Stopped: Funding unavailable
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2007NT031; WCC-52 (Other: Women's Cancer Center, University of Minnesota)
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Constipation; Bowel Obstruction; Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: constipation, impaction, and bowel obstruction; ovarian epithelial cancer; peritoneal cavity cancer; fallopian tube cancer
MeSH Terms: conditions — Constipation; Intestinal Obstruction; Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample (5 ml red top tube) will be drawn before the patient's first chemotherapy treatment, after the 3rd cycle of chemotherapy, at the post chemotherapy follow-up visit (approximately 30 days after chemotherapy is completed) and approximately 4 months after completion of chemotherapy at the time of a routine follow-up visit. Whenever possible, the blood will be drawn at the same time blood is being collected for clinical purposes therefore flexibility is allowed in the timing of the research related bloods.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients Receiving Chemotherapy: Patients with newly diagnosed ovarian, fallopian tube or primary peritoneal cancer for which 6 cycles of a taxane and platinum containing regimen is planned

SUMMARY:
RATIONALE: Gathering information about changes in serotonin levels in patients undergoing chemotherapy for ovarian cancer, fallopian tube cancer, or primary peritoneal cancer may help doctors learn more about constipation caused by chemotherapy.

PURPOSE: This clinical trial is studying how blood levels of serotonin effect constipation caused by chemotherapy in patients with newly diagnosed ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if there are any alterations in serotonin levels in patients undergoing chemotherapy for ovarian, fallopian tube, or primary peritoneal cancer and if this is associated with increased constipation.

OUTLINE: Patients undergo blood sample collection prior to beginning of planned postoperative chemotherapy, after 3 and 6 courses of chemotherapy, and at the 3-month surveillance visit. Patients also complete a bowel function questionnaire at these time points.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ovarian, fallopian tube, or primary peritoneal cancer
* Planned to undergo 6 courses of a taxane and platinum-containing regimen

Exclusion Criteria:

* Ovarian low malignant potential tumor
* History of constipation or irritable bowel syndrome
* History of colorectal cancer
* Prior bowel resection at time of staging/cytoreductive surgery
* Prior abdominal-pelvic radiation
* Prior bowel surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with newly diagnosed ovarian, fallopian tube, or primary peritoneal cancer.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Alterations in serotonin levels associated with increased constipation | PreDose, Post 3rd Cycle, Post Treatment and 4 Months Post Treatment
  Once the blood is drawn at the time of another necessary blood draw, the specimen will be labeled as a send out lab in the acute care lab. These are frozen and batched. Batched samples will then be sent to an outside laboratory for serotonin measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A. Geller, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States